CLINICAL TRIAL: NCT01396954
Title: Prevalence and Clinical Characteristics of the Patients With Liver Cirrhosis and Different Glucose Metabolism Disorders - A Prospective Study.
Brief Title: Cirrhosis-Diabetes
Acronym: CH-DM
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Hospital Universitario Dr. Jose E. Gonzalez (Other)
Responsible Party: Diego Garcia-Compean, Gastroenterology Service and Department of Internal Medicine, University Hospital
Other Study IDs: CREED-ENDO
Record Dates: First submitted 2011-07-18; First posted 2011-07-19 (Estimated); Last update posted 2011-07-19 (Estimated); Status verified 2007-11

CONDITIONS: Glucose Metabolism Disorders
Keywords: Liver cirrhosis; Diabetes mellitus; Hepatogenous diabetes; Oral glucose tolerance test; Insulin resistance.
MeSH Terms: conditions — Glucose Metabolism Disorders; Liver Cirrhosis; Diabetes Mellitus; Insulin Resistance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Glucose metabolism disorders (GMD) can be present in an overt and a subclinical way. They have negative impact in survival of patients with liver cirrhosis (LC). Their prevalence has not been determined in compensated cirrhotic patients.

DETAILED DESCRIPTION:
Overt Diabetes Mellitus (DM) is observed in 21 to 40% of patients with liver cirrhosis (LC). There are two ways in which DM is related to LC: firstly, type 2 diabetes mellitus (T2DM), which has a genetic component and is often associated with metabolic syndrome (obesity, hypertriglyceridemia, and hypertension), causes chronic liver disease (steatosis, steatohepatitis, and LC Secondly, LC may cause impaired glucose tolerance (IGT) and DM. During the initial stages of LC these metabolic disorders are subclinical as can only be detected by an oral glucose tolerance test (OGTT). As liver disease progresses, DM becomes clinically evident.

Diabetes mellitus secondary to LC is known as "hepatogenous diabetes" (HD). Although it has been accepted that the LC is a diabetogenic condition, HD is not recognized by the American Diabetes Association and the WHO. Cirrhosis caused by alcohol, HCV, and hemochromatosis are more frequently associated to HD than other etiologies . It has been observed that HCV core protein induces insulin resistance (IR), steatosis, and DM regardless of body mass index (BMI). Patients with chronic alcoholism often have chronic pancreatic damage resulting in DM . In short, T2DM and HD have different etiology, but they seem to have similar pathophysiologic mechanisms for liver function deterioration. They increase the risk of complications and death.

In recent years, the incidence of obesity has increased alarmingly in the world, particularly in the Western countries . In Mexico, overweight and obesity, which are suffered by about 70% of the adult population are a serious public health problem,. This figure puts this country in second place in the world, behind only the United States of America. The incidence of T2DM and metabolic syndrome has increased rapidly in our country . They have became the most common causes of cryptogenic cirrhosis in Mexico. Many published studies, which have reviewed the prevalence of DM in cirrhotic patients, do not make a distinction between T2DM and HD; additionally, subclinical glucose metabolism disorders (GMD) are not routinely identified, so the magnitude of the problem has been underestimated. On the other hand, the clinical and biochemical features of cirrhotic patients with different GMD are not known at present. The clinical distinction of GMD may be useful for prognosis and therapeutic purposes. Based on the aforementioned, the objectives of the present study were: a) To establish the prevalence of clinical and subclinical forms of GMD (T2DM, HD, IGT) in a cohort of patients with compensated LC of diverse etiology; and b) To determine the clinical and biochemical characteristics of patient with these different GMD and to find whether there are significant differences among them..

ELIGIBILITY:
Inclusion Criteria:

* the presence of biopsy- or clinically diagnosed liver cirrhosis; clinically compensated cirrhosis; age above 18 years; and any sexExclusion Criteria:
* Patients with complications due to liver disease (such as hepatocellular carcinoma, alcoholic hepatitis, active gastrointestinal bleeding, hepatic encephalopathy, hepatorenal syndrome, and severe infection)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We prospectively included patients with compensated liver cirrhosis who were admitted in the Regional Center for the Study of Digestive Diseases and the Liver Unit of the University Hospital and Faculty of Medicine
Sampling Method: Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2007-11; Primary Completion 2011-08 (Estimated); Study Completion 2012-08 (Estimated)